CLINICAL TRIAL: NCT06976827
Title: Prise en Charge de la dénutrition en Sortie d'Hospitalisation Par Des diététiciennes et Des Enseignants en activité Physique adapté à Domicile : étude de faisabilité (DENUTADOM)
Brief Title: Management of Undernutrition on Discharge From Hospital by Dieticians and Physical Activity Teachers at Home
Acronym: DENUTADOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier Henri Mondor d'Aurillac (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RIPH2_VILANOVA_DENUTADOM; IDRCB : 2025-A00416-43 (Other: ANSM)
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Malnutrition Severe; Malnutrition; Moderate
Keywords: moderate malnutrition; severe malnutrition; ambulatory care; discharge from hospital
MeSH Terms: conditions — Malnutrition; Lymphoma, Follicular | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- After-hospital, care by a private dietician and a physical activity teacher (Experimental): For this study, there is only one arm. After hospital discharge, the patient will have multi-professional monitoring of his undernutrition: private dietician, adapted physical activity teacher and general practitioner.
  Interventions: Other: Dietary and physical activity monitoring during the 3-months post-hospitalization period

INTERVENTIONS:
Other: Dietary and physical activity monitoring during the 3-months post-hospitalization period — Three consultations with a private dietician, one consultation with the general practitioner, three months of APA monitoring

SUMMARY:
The DENUTADOM study is a single-center feasibility study. It is an interventional research project involving human subjects (RIPH2), which will lead to a change in the care and treatment of adult patients diagnosed as suffering from moderate to severe undernutrition during hospitalization. The aim of this study was to assess patient compliance with a new undernutrition management program (diet and physical activity) at discharge from hospital.

In this study, during hospitalization, patients may be included in the study if they meet the inclusion criteria. To this end, the physician will offer to participate in the study, and will provide the patient with an information document. If the patient agrees to take part, he or she will be included in the study after signing the consent form. Participation will last 3 months.

On inclusion, after seeing the physician, an adapted physical activity teacher (EAPA) and a hospital dietician will assess the patient's physical capacities and dietary needs, in order to draw up an adapted physical and dietary program. The CRA will assess the patient's quality of life using a questionnaire. When the patient is discharged, he will be given a notebook in which to keep track of appointments with healthcare professionals (GP, private dietician, EAPA). Patients are also asked to keep a record of their non-protocol care appointments and participation in physical activities.

After hospitalization, the patient will have to follow a multi-professional program: dietetic by a private dietician (at D3-J5, at 3 weeks and then at 6 weeks), medical by the general practitioner (at 1 month), and adapted physical activity by the EAPA (during 3 months).

At three months, the patient will be seen again by the hospital's health professionals. The investigating physician will reassess nutritional status, and the EAPA will reassess physical capacity. The patient will be asked to return his diary so that data can be collected. They will also be given a quality of life and satisfaction questionnaire to complete.

When all patients have completed their follow-up, a satisfaction questionnaire will be sent to each healthcare professional.

Currently, as part of standard care, , dietetics and physical rehabilitation are not reimbursed. As a result, although recommended, patients rarely benefit from a dietetic consultation and adapted physical activity follow-up following a diagnosis of undernutrition. We therefore hypothesize that early cooperative outpatient care, involving general practitioners, private dieticians and adapted physical activity teachers (EAPA), for adult patients diagnosed as moderately or severely malnourished during hospitalization will optimize the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderately or severely malnourished adult patient according to HAS diagnostic criteria: At least one phenotypic criterion: weight loss (> 5% in 1 month, > 10% in 6 months or relative to pre-disease weight), BMI < 18.5 in < 70 years or BMI < 22 in ≥ 70 years, reduced muscle mass and/or function AND At least one etiological criterion: reduction in food intake > 50% for > 7 days or > 14 days regardless of reduction, reduced absorption, aggressive situation with hypercatabolism
* Patient with an attending physician wishing to participate in the study
* Patient wishing to be followed by a private dietician participating in the study

Exclusion Criteria:

* Patients with cognitive disorders
* Patients with eating disorders
* Pregnant or breast-feeding patient
* Patient with an estimated life expectancy of less than 6 months (at investigator's discretion)
* Patient under legal protection
* Patient not affiliated to the social security system
* Patient who has not signed a free, written and informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate patient compliance with a new management program (dietetics and physical rehabilitation) for undernutrition on discharge from hospital | Only once, at the 3 months follow-up
  Assessment of patient compliance with the innovative program will be based on their participation in the various consultations under the protocol (medical, dietary, physical rehabilitation), as well as in their adapted physical activity program. The clinical research associate in charge of the study will collect these data from the data transmitted by the professionals in charge of the patient's follow-up (physician, dietician, EAPA), as well as from the follow-up booklet completed by the patient.
  Adherence will be measured by analyzing deviations from consultations and APA sessions scheduled as part of the protocol, by category:
  * Medical: 2 scheduled consultations (attending general practitioner + hospital physician)
  * Dietetics: 3 consultations planned
  * Adapted physical activity: number of sessions varies according to the program defined by the EAPA

SECONDARY OUTCOMES:
Evaluate the patient's grip strength during the study | Three times : At inclusion, at 1 month and 3 months after inclusion
  Grip strength will be assessed using the handgrip, enabling muscle strength to be measured in kg. The grip strength test will be performed according to the Southampton protocol.
Evaluate the speed of chair lifting during the study | Three times : At inclusion, at 1 month and 3 months after inclusion
  Chair-lifting speed is assessed by the 5 chair-lifts test. This is a benchmark test for assessing muscle strength.
Evaluate the walking speed during the study | Three times : At inclusion, at 1 month and 3 months after inclusion
  Walking speed is assessed by the 4-meter walking test (4MWT). Walking speed over 4 meters is assessed to the nearest 0.01 second using a stopwatch. The test will be carried out twice in succession, and the fastest walking speed, expressed in m/s, will be used.
Evaluate the patient's weight during the study | Three times : At inclusion, at 1 month and 3 months after inclusion
  Weight will be measured in kilograms. Weight measurements at D0 and M3 will be taken on the same model of scale. As weight measurement at M1 is carried out at the attending physician's, the scale used will be different from that used for the other two measurement points.
Evaluate the patient's nutrition status during the study | Twice : At inclusion and at 3 months after inclusion
  The status of "undernourished" / "not undernourished" will be determined on the basis of the definition given in the latest HAS recommendations (Diagnosis of undernutrition in children and adults - November 2019 and Diagnosis of undernutrition in people aged 70 and over - November 2021).
Evaluate the patient's biological parameters during the study : phosphorus, magnesium, potassium, calcemia, corrected calcemia and transferrin-binding capacity | Three times : At inclusion, at 1 month and 3 months after inclusion
  The results of these biological parameters prescribed as standard for monitoring undernutrition will be recorded during the three medical visits, if values are available. The unit of measurement for these blood parameters will be the mmol/L.
Evaluate the patient's biological parameters relating to liver activity during the study : ASAT, ALAT, PAL, gamma-GT | Three times : At inclusion, at 1 month and 3 months after inclusion
  The results of these biological parameters prescribed as standard for monitoring undernutrition will be recorded during the three medical visits, if values are available. The unit of measurement for these blood parameters will be the UI/L.
Evaluate the patient's biological parameters during the study : albumin, pre-albumin, CRP, ferritin | Three times : At inclusion, at 1 month and 3 months after inclusion
  The results of these biological parameters prescribed as standard for monitoring undernutrition will be recorded during the three medical visits, if values are available. The unit of measurement for these blood parameters will be the g/L.
Evaluate the patient's quality of life during the study by the EQ-5D-5L questionnaire. | Three times : At inclusion, at 1 month and 3 months after inclusion
  Patients' quality of life will be assessed using the EQ-5D-5L questionnaire at three medical visits. The EQ-5D-5L questionnaire consists of a descriptive section and a visual analog scale. The descriptive part comprises five dimensions: mobility, personal care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated by the patient according to 5 degrees: no problems, mild problems, moderate problems, severe problems and extreme problems. The visual scale is a vertical analog scale, with the ends labelled "the best health you can imagine" (score : 100) and "the worst health you can imagine" (score : 0). The difference in score between the baseline and the two follow-up visits will be measured.
Evaluate end-of-study re-hospitalization and mortality rates | Only once, at the 3 months follow-up
  The number of re-hospitalized and deceased patients will be collected by the CRA from the patient's medical file and after discussion with the healthcare professionals in charge of the patient's follow-up.
Evaluate patient satisfaction with their care at the end of the study | Only once, at the 3 months follow-up
  It will be assessed using a 5-point satisfaction scale, from very dissatisfied to very satisfied.
At the end of the study, assess patients' consumption of out-of-protocol care | Only once, at the 3 months follow-up
  The use of dietary consultations, out-of-protocol physical rehabilitation sessions and complementary general medical consultations will be recorded by the CRA using a follow-up booklet completed by the patient.
Evaluate the satisfaction of each professional involved (doctor, dietician, EAPA) in this protocol | Only once, at the study completion
  The satisfaction of each professional involved (doctor, dietician, EAPA) in this protocol for the early management of undernutrition will be assessed using a 5-point satisfaction scale, from very dissatisfied to very satisfied.
Evaluate the medico-economic relevance of this new pathway for the early management of undernutrition | Only once, at the 3 months follow-up
  A cost-utility analysis will be carried out from both a societal and a health insurance perspective, in order to measure the relevance of the allocative efficiency of expenditure at M3. Utility will be calculated in relation to quality of life as measured by the EQ-5D-5L. Costs will be calculated on the basis of the following data:
  * For direct medical and non-medical costs: cost of medical treatment, cost of consultations, cost of complementary biological and radiological examinations, cost of medical transport and out-of-pocket expenses for patients;
  * For indirect costs: daily benefits related to work stoppage;
  * For intangible costs: psychological consequences of illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Henri Mondor d'Aurillac, Aurillac, France